CLINICAL TRIAL: NCT03246321
Title: Repetitive Electrostatic Pressurised Intraperitoneal Aerosol Chemotherapy With Oxaliplatin (ePIPAC-OX) as a Palliative Monotherapy for Isolated Unresectable Colorectal Peritoneal Metastases: Protocol of a Multicentre, Open-label, Single-arm, Phase II Study (CRC-PIPAC)
Brief Title: PIPAC for Peritoneal Metastases of Colorectal Cancer
Acronym: CRC-PIPAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Koen Rovers (Other)
Responsible Party: Sponsor-Investigator, Koen Rovers, MD, Coordinating Investigator, Catharina Ziekenhuis Eindhoven
Organization: Catharina Ziekenhuis Eindhoven (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL60405.100.17; 2017-000927-29 (EudraCT Number); NTR6603 (Registry Identifier: NTR); ISRCTN89947480 (Registry Identifier: ISRCTN); NL60405.100.17 (Other: Dutch Competent Authority)
Record Dates: First submitted 2017-08-02; First posted 2017-08-11 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Colorectal Neoplasms; Peritoneal Neoplasms; Appendiceal Neoplasms; Peritoneal Carcinomatosis
Keywords: Colorectal Neoplasms; Peritoneal Neoplasms; Intraperitoneal Injections; Laparoscopy; Aerosols; Chemotherapy, Cancer, Regional Perfusion; Antineoplastic Agents; Leucovorin; Fluorouracil; Platinum; Intraoperative Complications; Postoperative Complications; Drug-Related Side Effects and Adverse Reactions; Disease-free survival; Survival; Mortality; Quality of Life; Costs and Cost Analysis; Translational Medical Research; Clinical Trials, Phase II as topic; PIPAC; Pressurized Intraperitoneal Aerosol Chemotherapy; Pressurised Intraperitoneal Aerosol Chemotherapy; Peritoneum; Cecal Neoplasms; Oxaliplatin
MeSH Terms: conditions — Colorectal Neoplasms; Peritoneal Neoplasms; Appendiceal Neoplasms; Neoplasms; Intraoperative Complications; Postoperative Complications; Drug-Related Side Effects and Adverse Reactions; Cecal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- repetitive ePIPAC-OX (Experimental)
  Interventions: Combination Product: repetitive ePIPAC-OX

INTERVENTIONS:
Combination Product: repetitive ePIPAC-OX — Instead of standard palliative treatment, enrolled patients receive laparoscopy-controlled electrostatic pressurised intraperitoneal aerosol chemotherapy with oxaliplatin (ePIPAC-OX) (92 mg/m2 body-surface area [BSA]) with intravenous leucovorin (20 mg/m2 BSA) and bolus 5-fluorouracil (400 mg/m2 BSA) every six weeks. Four weeks after each procedure, patients undergo clinical, radiological, and biochemical evaluation. ePIPAC-OX is repeated until clinical, radiological, or macroscopic disease progression, after which standard palliative treatment is (re)considered.

SUMMARY:
This is multicentre, open-label, single-arm phase II study that investigates the feasibility, safety, tolerability, preliminary efficacy, costs, and pharmacokinetics or repetitive electrostatic pressurised intraperitoneal aerosol chemotherapy (ePIPAC-OX) as a palliative monotherapy for patients with isolated unresectable colorectal peritoneal metastases.

DETAILED DESCRIPTION:
Rationale: repetitive electrostatic pressurised intraperitoneal aerosol chemotherapy with oxaliplatin (ePIPAC-OX) is offered as a palliative treatment option for patients with isolated unresectable colorectal peritoneal metastases (PM) in several centres worldwide. However, little is known about its feasibility, safety, tolerability, efficacy, costs, and pharmacokinetics in this setting.

Objectives: to prospectively explore the feasibility, safety, tolerability, preliminary efficacy, costs, and pharmacokinetic profile of repetitive ePIPAC-OX as a palliative monotherapy for isolated unresectable colorectal PM under controlled circumstances.

Study design: multicentre, open-label, single-arm, phase II study.

Setting: two Dutch tertiary referral hospitals for the surgical treatment of colorectal PM.

Study population: adults who have a World Health Organisation (WHO) performance status of 0 or 1, adequate organ functions, histologically or cytologically confirmed unresectable PM of a colorectal or appendiceal carcinoma, no systemic metastases, no symptoms of gastrointestinal obstruction, no contraindications for the planned intervention, and no previous pressurised intraperitoneal aerosol chemotherapy (PIPAC).

Intervention: instead of standard palliative treatment, enrolled patients receive laparoscopy-controlled ePIPAC-OX (92 mg/m2 body-surface area [BSA]) with intravenous leucovorin (20 mg/m2 BSA) and bolus 5-fluorouracil (400 mg/m2 BSA) every six weeks. Four weeks after each procedure, patients undergo clinical, radiological, and biochemical evaluation. ePIPAC-OX is repeated until clinical, radiological, or macroscopic disease progression, after which standard palliative treatment is (re)introduced.

Outcomes: the primary outcome is the number of patients with major toxicity (grade ≥3 according to the Common Terminology Criteria for Adverse Events v4.0) up to four weeks after the last procedure. Secondary outcomes are the environmental safety of ePIPAC-OX, procedure-related characteristics, the number of procedures in each patient and reasons for discontinuation, minor toxicity, organ-specific toxicity, postoperative complications, hospital stay, readmissions, quality of life, costs, progression-free survival, overall survival, and the radiological, histopathological, cytological, biochemical, and macroscopic tumour response. Atomic absorption spectrophotometry is used to measure concentrations of oxaliplatin in plasma, plasma ultrafiltrate, urine, ascites, PM, and normal peritoneum during and after ePIPAC-OX.

ELIGIBILITY:
Eligible patients are adults who have:

* a World Health Organisation (WHO) performance status of ≤1;
* histological or cytological proof of PM of a colorectal or appendiceal carcinoma;
* unresectable disease determined by abdominal computed tomography (CT) and a diagnostic laparoscopy or laparotomy;
* adequate organ functions (haemoglobin ≥5.0 mmol/L, neutrophils ≥1.5 x 109/L, platelets ≥100 x 109/L, serum creatinine <1.5 x ULN, creatinine clearance ≥30 ml/min, and liver transaminases <5 x ULN);
* no symptoms of gastrointestinal obstruction;
* no radiological evidence of systemic metastases;
* no contraindications for oxaliplatin or 5-fluorouracil/leucovorin;
* no contraindications for a laparoscopy;
* no previous PIPAC-procedures.

Enrolled patients are excluded from the analyses in case they did not receive a first ePIPAC-OX, e.g.:

* due to systemic metastases on baseline thoracoabdominal CT, or;
* due to non-access during first ePIPAC-OX, or;
* due to resectable disease during first ePIPAC-OX.

Importantly, enrolment is allowed for patients with an unresected primary tumour (if asymptomatic) and for patients in various lines of palliative treatment, including patients who refuse, have not had, or do not qualify for first-line palliative systemic therapy. All potentially eligible patients are discussed by a multidisciplinary team. Enrolled patients are informed about the potential consequences of postponing or discontinuing standard palliative treatment by a medical oncologist prior to enrolment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Major toxicity | Expected (in case of three ePIPAC-OX): 16 weeks
  Number of patients with Common Terminology Criteria for Adverse Events (CTCAE) v4.0 grade III-V, up to 4 weeks after the last ePIPAC-OX

SECONDARY OUTCOMES:
Minor toxicity | Expected (in case of three ePIPAC-OX): 16 weeks
  Number of patients with Common Terminology Criteria for Adverse Events (CTCAE) v4.0 grade II, up to 4 weeks after the last ePIPAC-OX
Organ-specific toxicity | Expected (in case of three ePIPAC-OX): 16 weeks
  Number of patients that develops bone marrow, kidney, or liver function disorders, up to four weeks after the last ePIPAC-OX
Major postoperative complications | Expected (in case of three ePIPAC-OX): 16 weeks
  Number of patients with Clavien-Dindo grade III-V postoperative complications, up to four weeks after the last ePIPAC
Minor postoperative complications | Expected (in case of three ePIPAC-OX): 16 weeks
  Number of patients with Clavien-Dindo grade II postoperative complications, up to four weeks after the last ePIPAC-OX
Hospital stay | Expected (in case of three ePIPAC-OX): 16 weeks
  Number of days between ePIPAC-OX and initial discharge, up to four weeks after the last ePIPAC-OX
Readmissions | Expected (in case of three ePIPAC-OX): 16 weeks
  Number of hospital admissions after initial discharge after ePIPAC-OX, up to four weeks after the last ePIPAC-OX
Radiological tumour response | Expected (in case of three ePIPAC-OX): 16 weeks
  Number of patients with radiological response/stable disease/progression, based on central review of thoracoabdominal CT and diffusion-weighted MRI at baseline and four weeks after each ePIPAC-OX, performed by two independent radiologists blinded to clinical outcomes (classification not defined a priori)
Histopathological tumour response | Expected (in case of three ePIPAC-OX): 12 weeks
  Peritoneal Regression Grading Score (PRGS), based on central review of collected peritoneal biopsies during each ePIPAC-OX, performed by two independent pathologists blinded to clinical outcomes
Cytological tumour response | Expected (in case of three ePIPAC-OX): 12 weeks
  Number of patients with positive/negative cytology, based on collected ascites or peritoneal washing cytology during each ePIPAC-OX
Macroscopic tumour response | Expected (in case of three ePIPAC-OX): 12 weeks
  Peritoneal Cancer Index and ascites volume during each ePIPAC-OX
Biochemical tumour response | Expected (in case of three ePIPAC-OX): 16 weeks
  Tumour marker value measured at baseline, each postoperative day, and four weeks after each ePIPAC-OX
Quality of life: EQ-5D-5L | Expected (in case of three ePIPAC-OX): 16 weeks
  EQ-5D-5L at baseline and one and four weeks after each ePIPAC-OX
Quality of life: QLQ-C30 | Expected (in case of three ePIPAC-OX): 16 weeks
  QLQ-C30 at baseline and one and four weeks after each ePIPAC-OX
Quality of life: QLQ-CR29 | Expected (in case of three ePIPAC-OX): 16 weeks
  QLQ-CR29 at baseline and one and four weeks after each ePIPAC-OX
Costs | Expected (in case of three ePIPAC-OX): 16 weeks
  Costs of treatment, based on questionnaires (iMTA PCQ, iMTA MCQ) four weeks after each ePIPAC-OX, derived from the Dutch costing guidelines for health care research at the time of analysis
Progression-free survival | 24 months
  Time between enrolment and clinical, radiological, or macroscopic progression, or death
Overall survival | 24 months
  Time between enrolment and death
Environmental safety of ePIPAC-OX | 1 week (measured only during the first three procedures in the study)
  Platinum concentrations in the air of the operating room and on the surface of the operating room during ePIPAC-OX
Pharmacokinetics | Expected (in case of three ePIPAC-OX): 13 weeks
  Platinum concentrations in plasma and plasma ultrafiltrate (collected before ePIPAC-OX and 5, 10, 20, 30, 60, 120, 240, 360, and 1080 minutes after oxaliplatin injection), urine (collected before ePIPAC-OX and on postoperative days 1, 3, 5, and 7), and two pieces of normal peritoneum and two peritoneal metastases collected during each ePIPAC-OX.
Procedure-related characteristics: intraoperative complications | Expected (in case of three ePIPAC-OX): 12 weeks
  Number of procedures with intraoperative complications determined during each ePIPAC-OX
Procedure-related characteristics: adhesions | Expected (in case of three ePIPAC-OX): 12 weeks
  Zühlke score determined during each ePIPAC-OX
Procedure-related characteristics: operating time | Expected (in case of three ePIPAC-OX): 12 weeks
  Operating time in minutes determined during each ePIPAC-OX
Procedure-related characteristics: blood loss | Expected (in case of three ePIPAC-OX): 12 weeks
  Blood loss in minutes determined during each ePIPAC-OX

CONTACTS AND LOCATIONS:
Overall Officials: Ignace de Hingh, MD, PhD, Study Chair — Catharina Hospital, Eindhoven, Netherlands; Djamila Boerma, MD, PhD, Principal Investigator — St Antonius Hospital, Nieuwegein, Netherlands
Locations (2):
- Netherlands (2):
  - Catharina Hospital, Eindhoven
  - St. Antonius Hospital, Nieuwegein

IPD SHARING:
Plan to Share IPD: Yes
Available on request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: End of the study
Access Criteria: Available on request

REFERENCES:
- [Background] Giger-Pabst U, Tempfer CB. How to Perform Safe and Technically Optimized Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC): Experience After a Consecutive Series of 1200 Procedures. J Gastrointest Surg. 2018 Dec;22(12):2187-2193. doi: 10.1007/s11605-018-3916-5. Epub 2018 Aug 21. PMID 30132291
- [Background] Tempfer C, Giger-Pabst U, Hilal Z, Dogan A, Rezniczek GA. Pressurized intraperitoneal aerosol chemotherapy (PIPAC) for peritoneal carcinomatosis: systematic review of clinical and experimental evidence with special emphasis on ovarian cancer. Arch Gynecol Obstet. 2018 Aug;298(2):243-257. doi: 10.1007/s00404-018-4784-7. Epub 2018 Jun 4. PMID 29869089
- [Background] Grass F, Vuagniaux A, Teixeira-Farinha H, Lehmann K, Demartines N, Hubner M. Systematic review of pressurized intraperitoneal aerosol chemotherapy for the treatment of advanced peritoneal carcinomatosis. Br J Surg. 2017 May;104(6):669-678. doi: 10.1002/bjs.10521. PMID 28407227
- [Derived] van de Vlasakker VCJ, Lurvink RJ, Wassenaar EC, Rauwerdink P, Bakkers C, Rovers KP, Bonhof CS, Burger JWA, Wiezer MJ, Boerma D, Nienhuijs SW, Mols F, de Hingh IHJT. Comparing patient reported abdominal pain between patients treated with oxaliplatin-based pressurized intraperitoneal aerosol chemotherapy (PIPAC-OX) and primary colorectal cancer surgery. Sci Rep. 2023 Nov 22;13(1):20458. doi: 10.1038/s41598-023-47510-0. PMID 37993560
- [Derived] Lurvink RJ, Rovers KP, Wassenaar ECE, Bakkers C, Burger JWA, Creemers GM, Los M, Mols F, Wiezer MJ, Nienhuijs SW, Boerma D, de Hingh IHJT. Patient-reported outcomes during repetitive oxaliplatin-based pressurized intraperitoneal aerosol chemotherapy for isolated unresectable colorectal peritoneal metastases in a multicenter, single-arm, phase 2 trial (CRC-PIPAC). Surg Endosc. 2022 Jun;36(6):4486-4498. doi: 10.1007/s00464-021-08802-6. Epub 2021 Nov 10. PMID 34757489
- [Derived] Rovers KP, Wassenaar ECE, Lurvink RJ, Creemers GM, Burger JWA, Los M, Huysentruyt CJR, van Lijnschoten G, Nederend J, Lahaye MJ, Deenen MJ, Wiezer MJ, Nienhuijs SW, Boerma D, de Hingh IHJT. Pressurized Intraperitoneal Aerosol Chemotherapy (Oxaliplatin) for Unresectable Colorectal Peritoneal Metastases: A Multicenter, Single-Arm, Phase II Trial (CRC-PIPAC). Ann Surg Oncol. 2021 Sep;28(9):5311-5326. doi: 10.1245/s10434-020-09558-4. Epub 2021 Feb 5. PMID 33544279
- [Derived] Lurvink RJ, Tajzai R, Rovers KP, Wassenaar ECE, Moes DAR, Pluimakers G, Boerma D, Burger JWA, Nienhuijs SW, de Hingh IHJT, Deenen MJ. Systemic Pharmacokinetics of Oxaliplatin After Intraperitoneal Administration by Electrostatic Pressurized Intraperitoneal Aerosol Chemotherapy (ePIPAC) in Patients with Unresectable Colorectal Peritoneal Metastases in the CRC-PIPAC Trial. Ann Surg Oncol. 2021 Jan;28(1):265-272. doi: 10.1245/s10434-020-08743-9. Epub 2020 Jun 22. PMID 32572849
- [Derived] Rovers KP, Lurvink RJ, Wassenaar EC, Kootstra TJ, Scholten HJ, Tajzai R, Deenen MJ, Nederend J, Lahaye MJ, Huysentruyt CJ, van 't Erve I, Fijneman RJ, Constantinides A, Kranenburg O, Los M, Thijs AM, Creemers GM, Burger JW, Wiezer MJ, Boerma D, Nienhuijs SW, de Hingh IH. Repetitive electrostatic pressurised intraperitoneal aerosol chemotherapy (ePIPAC) with oxaliplatin as a palliative monotherapy for isolated unresectable colorectal peritoneal metastases: protocol of a Dutch, multicentre, open-label, single-arm, phase II study (CRC-PIPAC). BMJ Open. 2019 Jul 27;9(7):e030408. doi: 10.1136/bmjopen-2019-030408. PMID 31352425